CLINICAL TRIAL: NCT06878885
Title: Trauma and Cardiometabolic Health in an American Indian Community
Acronym: IHPIPO'TO'TSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Baylor University (Other); Blackfeet Community College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 163237; 5R01HL163237-02 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Psychological Stress; Cardiometabolic Conditions; Mental Health
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study is designed to examine cardiovascular, neuroendocrine, and inflammatory responses to a brief (4 minutes) mental arithmetic task (i.e., a psychological challenge) in the laboratory. Cardiovascular activity will be measured during a resting baseline period (10 minutes) and during the task (4 minutes). Participants will provide salivary samples before the task and after the task (~20-90 minutes) which will be used to assess neuroendocrine (i.e., cortisol) and inflammatory (i.e., IL-6). Cardiovascular, neuroendocrine, and inflammatory responses will be examined in relation to other study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paced Auditory Serial Addition Task (Experimental): Volunteers are presented with an audio playing of single digit numbers between 1 and 9. They are instructed to add the number with the number previously presented and say the answer out loud. Volunteers are told their performance is being scored by research assistants. Volunteers are also instructed to look at themselves in a mirror while partaking in the task. Volunteers are informed they can discontinue at any time. Volunteers complete brief questionnaires before and after the task to asses their perceptions of stress, arousal, and anxiety.
  Interventions: Behavioral: Acute psychological stress task (Paced Auditory Serial Addition Task)

INTERVENTIONS:
Behavioral: Acute psychological stress task (Paced Auditory Serial Addition Task) — Volunteers will complete a 4-minute Paced Auditory Serial Addition Task which is a standardized laboratory challenge that is widely used to monitor cardiovascular, neuroendocrine, and inflammatory responses in the laboratory.

SUMMARY:
Volunteers for the study are asked to participate in two laboratory sessions. In the first laboratory session, volunteers are asked to provide a blood sample which will be used to measure factors related to health. Participants also complete questionnaires related to demographic and health-related information and undergo evaluations of their body composition. In the second laboratory visit, participants are asked to have cardiovascular, neuroendocrine, and inflammatory activity measured during a brief period of rest and during a short challenging psychological task. Participants will also complete questionnaires. The study is designed to examine the associations between experiences such as trauma and resiliency with changes in bodily systems during a challenge and current health.

DETAILED DESCRIPTION:
This cross-sectional study will examine the association between factors of resiliency and trauma with physiological (cardiovascular, neuroendocrine, inflammatory) responses to acute stress and current mental and physical health. Study volunteers will include individuals who identify as American Indian and currently live on and near the Blackfeet Reservation. Study volunteers will be asked to provide information that will be used to measure: correlates of cardiometabolic and mental health, acute psychological stress, arterial stiffness. Results of the study will help increase knowledge of cardiometabolic and mental health in the context of past and ongoing trauma and resiliency.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Identifying as American Indian
* Living on or near Blackfeet reservation

Exclusion Criteria:

* Uncontrolled hypertension

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in systolic blood pressure activity from baseline to task | 10 minute resting baseline mean will be subtracted from the 4 minute task period for each value
  The mean systolic blood pressure (mmHg) will be subtracted from the mean of the task period.
Changes in diastolic blood pressure activity from baseline to task | 10 minute resting baseline mean will be subtracted from the 4 minute task period for each value
  The mean diastolic blood pressure (mmHg) will be subtracted from the mean of the task period.
Changes in heart rate activity from baseline to task | 10 minute resting baseline mean will be subtracted from the 4 minute task period for each value
  The mean heart rate (bpm) will be subtracted from the mean of the task period.
Change in cortisol from baseline to task | Baseline will be subtracted from the peak (15 minutes after task onset, 35 minute task onset)
  Salivary samples will be taken to measure cortisol (nmol/L) the mean from the peak stress period will be subtracted from the baseline
Changes in IL-6 from baseline to task | Baseline will be subtracted from the level 30 minutes after task onset.
  IL-6 (pg/mL) measured at baseline will be subtracted from the IL-6 measured post task.
Pulse wave velocity | 5 minutes
  Pulse wave velocity in m/s will be assessed by dual impedance cardiography as a non-invasive indicator of arterial stiffness. This measure will be derived from the 5 minute baseline period.
Resting systolic blood pressure | 10 minutes
  Resting systolic blood pressure (mmHg)
Resting diastolic blood pressure | 10 minutes
  Resting diastolic blood pressure (mmHg)
Inflammatory and anti-inflammatory cytokines | 5 minutes
  Circulating levels of C-reactive protein, interleukin-6, tumor necrosis factor-a, monocyte chemoattractant protein-1, interleukin-1b, interleukin-10, and adiponectin will be assessed via a blood draw. A composite score will be created.
Hemoglobin A1c | 5 minutes
  Hemoglobin A1c (nmol/L) will be assessed via blood draw
Glucose | 5 minutes
  Glucose (nmol/L) will be assessed via blood draw
Insulin | 5 minutes
  Insulin (mL) will be assessed via blood draw
Cholesterol | 5 minutes
  Total cholesterol (mg) will be assessed via blood draw
Low-density lipoprotein | 5 minutes
  Low-density lipoprotein (mg/dL) will be assessed via blood draw
High-density lipoprotein | 5 minutes
  high-density lipoprotein (mg/dL) will be assessed via blood draw
Triglycerides | 5 minutes
  Triglycerides (mmol/L) will be assessed via blood draw
Waist circumference | 2 minutes
  Waist circumference
Hip circumference | 2 minutes
  Hip circumference
Depressive symptomology (Hospital Anxiety Depression Questionnaire depression subscale) | 10 minutes
  Hospital Anxiety Depression Questionnaire (depression subscale)
Depressive symptomology (PHQ-9) | 10 minutes
  PHQ-9
Anxiety symptomtology | 5 minutes
  Hospital Anxiety Depression Questionnaire (Anxiety subscale)
Alcohol use | 10 minutes
  Alcohol use will be assessed using the Alcohol Use Identification Test
Substance use | 5 minutes
  A cumulative score of substance use will be reported by indicating the number of recreational drugs "ever" tried

CONTACTS AND LOCATIONS:
Overall Officials: Neha John-Henderson, PhD, Principal Investigator — Montana State University; Annie Ginty, PhD, Principal Investigator — Baylor University; Betty Henderson-Mathews, MA, Principal Investigator — Blackfeet Community College
Locations (1):
- Blackfeet Community College, Browning, Montana, United States